CLINICAL TRIAL: NCT07180862
Title: A Phase 1, Randomized, Double-blind Study to Compare the Pharmacokinetics, Between BAT3306 and Keytruda® (Pembrolizumab) in Participants With Stage IB-IIIA Non-small Cell Lung Cancer Following Complete Resection
Brief Title: A Study Evaluating BAT3306 Compared With Keytruda® in NSCLC Cancer Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BAT-3306-003-CR
Record Dates: First submitted 2025-08-19; First posted 2025-09-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: double-blind, randomized
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAT3306 (Experimental): Once every 3 weeks for a maximum of 1 year (not exceeding 18 cycles).
  Interventions: Drug: BAT3306
- US-Keytruda® arm (Active Comparator): Once every 3 weeks for a maximum of 1 year (not exceeding 18 cycles).
  Interventions: Drug: US-Keytruda®

INTERVENTIONS:
Drug: BAT3306 — One vial of 4 mL of concentrate contains 100 mg of BAT3306
  Other Names: Pembrolizumab Injection
  Arms: BAT3306
Drug: US-Keytruda® — One vial of 4 mL of concentrate contains 100 mg of pembrolizumab
  Other Names: Pembrolizumab Injection
  Arms: US-Keytruda® arm

SUMMARY:
Comparing the PK similarity of BAT3306 and Keytruda; in NSCLC participants who were completely removed by surgery as an auxiliary treatment

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-controlled, Phase 1 clinical study to evaluate the PK similarity of BAT3306 versus Keytruda® as adjuvant therapy in participants with early stage NSCLC. Participants must have no EGFR gene mutation or ALK gene rearrangement, have not received neoadjuvant or adjuvant radiotherapy and/or neoadjuvant chemotherapy, and have no plans for such treatment. A total of approximately 140 eligible participants will be randomly assigned in a 1:1 ratio to 2 double-blind treatment groups.

Participants who meet all inclusion criteria and none of exclusion criteria will be randomized in an Interactive Web Response System (IWRS).

All participants will receive the investigational medicinal product at 200 mg via intravenous infusion every 3 weeks for a treatment period of up to 12 months . Serum samples will be collected from participants at specified time points for PK analysis to evaluate the PK similarity and PK characteristics of BAT3306 versus Keytruda®, while also assessing their immunogenicity and safety, and preliminarily comparing their improvement in disease-free survival (DFS).

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria:

  1. Male or female, aged ≥18 and ≤75 years on the day of signing the Informed Consent Form (ICF);
  2. Participants are able to give voluntary informed consent and understand the study and are willing to follow and complete all the test procedures;
  3. Pathologically confirmed non-small cell lung cancer (NSCLC) after surgery, with a clear histological type and a pathology report provided;

Exclusion Criteria:

* Participants who meet any of the following criteria will be excluded from the study:

  1. Presence of EGFR gene mutation;
  2. Pathological diagnosis of small cell lung cancer or mixed tumors with small cell components, large cell neuroendocrine carcinoma (LCNEC), or sarcomatoid tumors;
  3. Have previously received any of the following treatments:

     Have received > 4 cycles of adjuvant chemotherapy. Prior neoadjuvant therapy. Major surgery within 4 weeks prior to randomization (including surgery for the primary neoplasm, but excluding vascular access procedures), or expected to undergo major surgery during the study.

     Use of Chinese herbal medicine with anti-tumor indications within 14 days prior to randomization.

     Use of growth factor support therapy or have received a transfusion within 14 days prior to randomization.
  4. Prior treatment with anti-PD-1, anti-PD-L1/2, anti-CD137, CTLA-4 modulators, or any other immunomodulatory agents.
  5. Severe acute or chronic infection, including any active infection requiring systemic anti-infective therapy within 2 weeks prior to randomization;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
PK equivalence | Cycle 1 day 1, day 2, day 3, day 5, day 8, day 15, day 22(each cycle is 21 days)
  To compare the pharmacokinetic (PK) similarity of BAT3306 versus US-Keytruda® as adjuvant therapy in participants with completely resected NSCLC：AUC0-τ, ss

SECONDARY OUTCOMES:
PK equivalence | Cycle 1，2，3，4，5，6，8，12，18（each cycle is 21 days）
  To evaluate the PK characteristics of BAT3306 and US-Keytruda® in participants with completely resected NSCLC：Cthough
immunogenicity equivalence | Weeks 2, 4,12,18,24
  To evaluate the immunogenicity of BAT3306 and US-Keytruda® in participants with completely resected NSCLC:Anti-drug antibody (ADA) positive rate at Weeks 2, 4,12,18,24
Vital signs | The third week of every 4 cycles and EOT（No more than 18 cycles）（each cycle is 21 days)
  Number of cases with abnormal vital signs results
Physical examination | The third week of every 4 cycles and EOT（No more than 18 cycles）（each cycle is 21 days)
  Number of cases with abnormal Physical examination results
Laboratory Examination | The third and sixth weeks of every 4 cycles and EOT（No more than 18 cycles）（each cycle is 21 days)
  Number of cases with abnormal Laboratory Examination results
Adverse event | The third week of every 4 cycles and EOT（No more than 18 cycles）（each cycle is 21 days)
  Number of cases with all adverse medical events that occur after the subject receives the investigational drug assessed by CTCAE V5.0
DFS（Disease-free survival） | Through study completion, No more than of 1 year
  the duration of the absence of tumor recurrence or metastasis as per the RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Dong, Dr., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science & Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No